CLINICAL TRIAL: NCT00320931
Title: Assessment of Coronary Flow Reserve and CT Angiography By Hybrid PET/CT: Relation to Clinically Indicated SPECT Studies
Brief Title: Assessment of Coronary Artery Disease by Hybrid PET/CT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Vasken Dilsizian, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-27314 (LR-05-003)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; PET CT scan; Stress test; Rubidium
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hybrid PET/CT (Experimental)
  Interventions: Device: Hybrid PET/CT

INTERVENTIONS:
Device: Hybrid PET/CT — Rest and vasodilation stress rubidium PET and coronary angiography with CT were performed using standard doses for clinically indicated studies.
  Other Names: Philips Gemini

SUMMARY:
There have been many advances in the test used to look for heart disease. An example of this newer technology is the Multislice CT scan (MSCT) and Positron Emission Tomography (PET) scans.

The use of this type of combined scan may show early coronary artery disease or the degree of damaged heart muscle form a heart attack with a single exam. It may help doctors to know who might benefit from heart surgery or angioplasty to increase the blood flow to the heart. This type of detailed images has previously been available only through cardiac catheterization.

DETAILED DESCRIPTION:
Advances in Non-invasive Multislice CT Imaging: Multislice CT (MSCT) and PET imaging are becoming more widely available and more useful in cardiac assessment. MSCT provides quantification of coronary calcium as well as information about the structures of the coronary vessel walls and atherosclerotic plaques. Multiple studies have demonstrated that MSCT provides information on coronary artery stenosis comparable to that obtained from invasive coronary angiography. PET imaging provides functional data via the measurement of coronary flow reserve (CFR). CFR is a quantitative measure of the increase in coronary blood flow in response to vasodilation; normal coronary flow is able to augment by three- to four-fold; diseased coronary arteries show less ability to increase flow, i.e. less CFR. Assessment of CFR yields functional information about the significance of coronary disease and is often used clinically in conjunction with anatomic imaging to identify early atherosclerosis. There is no current data evaluating the incremental value of hybrid PET/CT assessment of CFR and coronary anatomy in relation to SPECT studies in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older and able to give informed consent.
* Scheduled for clinically indicated gated Adenoscan SPECT studies at the University of Maryland Medical Center or Baltimore VA Center
* Documentation from participant's health care provider indicating no objection to subject's participation in study.

Exclusion Criteria:

* Hepatic; thyroid or renal disease (creatinine >1.5 or GFR < 60mL/min)
* Women of childbearing age not using medically acceptable form of contraception, pregnant or breast-feeding
* Contrast allergy
* Inability to cooperate with imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasken Dilsizian, M.D., Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 2006 to 2008 at the University of Maryland Medical Center
Pre-assignment Details: Enrolled participants who were claustrophobic did not complete the studies
Groups:
- Hybrid PET/CT: The participants underwent rest and vasodilator rubidium PET and CT angiography studies using standard doses for clinically indicated studies
Period: Overall Study
Arm/Group | Hybrid PET/CT
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Undergoing Imaging Studies
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: over 18 years] | 30 [19 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: The Incremental Value of Adenosine Flow Reserve by Rubidium PET to Clinically Acquired Gated Studies.
Description: All data were acquired in list-mode for 8 minutes and retrospectively sorted into static, ECG gated and dynamic images. Rubidium retention was calculated by dividing the late (3-8 minute) whole myocardium region-of-interest data by the integral of the input function over the first minute. Adenosine flow reserve was estimated by dividing rubidium retention during adenosine vasodilation by the same measure at rest. These quantitative flow and flow reserve values were compared to clinically acquired gated studies in the 30 participants.
Time Frame: 3-8 minute
Population: This study was terminated and the hybrid PET/CT scanner that was available to use for the study at the University of Maryland Medical Center was unable to generate quantitatively accurate absolute myocardial blood flow values. As such, we were unable to have scientifically accurate results and data to report.
Arm/Group | Subjects Undergoing Imaging Studies
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Subjects Undergoing Imaging Studies
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
For rubidium PET, statistical noise in static or gated images and quantitative accuracy in early-phase dynamic images could not be simultaneously optimized on the hybrid PET/CT scanner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No